CLINICAL TRIAL: NCT03880318
Title: Joint Preserving Surgery for Correction of Spasmodic Flat- Foot in Skeletally Mature Foot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Bahy Abdelaziz Ahmed, resident at Assiut University hospitals, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: spasmodic flat foot
Record Dates: First submitted 2018-12-30; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Flat Foot; Rigid; Flat Foot; Spastic
MeSH Terms: conditions — Flatfoot; Muscle Rigidity; Muscle Spasticity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- spasmodic flat foot (Other): extensor digitorum longus, peroneus brevis and tertius lengthening together with calcaneal osteotomies in spasmodic flat foot
  Interventions: Procedure: Joint Preserving Surgery in spasmodic flat foot

INTERVENTIONS:
Procedure: Joint Preserving Surgery in spasmodic flat foot — extensor digitorum longus, peroneus brevis and tertius lengthening together with calcaneal osteotomies

SUMMARY:
the investigators want to obtain a functional and radiological outcome of peroneus brevis, tertius and extensor digitorum longus muscles lengthening together with calcaneal osteotomies in the treatment of the spasmodic flat- foot.

DETAILED DESCRIPTION:
One of the most common foot complaints is the "flatfoot" deformity. Clinical evaluation of flatfeet primarily focuses on differentiation between the two main types: flexible and rigid. The rigid flatfoot deformity is an uncommon diagnosis (occurring one-third as often as the flexible type) but often is symptomatic and requires treatment". Multiple causes of rigid flatfeet have been identified such as rheumatoid arthritis, tarsal coalitions (being the most common cause) that are excluded from that research. Triple arthrodesis is used for treatment of rigid flat foot but the patient satisfaction is not good as there is some stiffness in the foot .but here the investigators want to know what is the effect of extensor digitorum longus, peroneus brevis and tertius lengthening together with osteotomies in alignment of spasmodic flat- foot. In patient with rigid flat- foot or spasmodic flat- foot will often have the hind-foot alignment to the outside. Alignment of the heel influences how weight-bearing stress is applied to the foot, ankle, knee and hip. So, these patients may benefit from the calcaneal osteotomies and extensor digitorum longus, peroneus brevis and tertius lengthening to improve that alignment.

ELIGIBILITY:
Inclusion Criteria:

* Painful, incorrectable pes Plano valgus after failure of conservative treatment
* Age: patients with skeletally mature foot as proved by x-ray

Exclusion Criteria:

* coalition bar
* Ankle subtalar joint arthritis.
* Previous foot fractures.
* Severe trophic skin disorders
* Standard contraindications to any surgery such as poor circulation, concurrent infection, other co-morbidity".

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
assess the foot deformity | Baseline
  assess foot deformity : full correction (valgus<10 degree), partial correction(valgus<15 degree),valgus >15 degree)
assess the pain: Visual Analog Score | Baseline
  The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. This tool was first used in psychology by Freyd in 1923